CLINICAL TRIAL: NCT02634853
Title: A Safety and Efficacy Study of Tavilermide Ophthalmic Solution for the Treatment of Dry Eye
Brief Title: A Safety and Efficacy Study of Tavilermide (MIM-D3) Ophthalmic Solution for the Treatment of Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mimetogen Pharmaceuticals USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIM-727
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Dry Eye
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tavilermide Ophthalmic Solution (Active Comparator): 1% Tavilermide Ophthalmic Solution
  Interventions: Drug: 1% Tavilermide Ophthalmic Solution
- Vehicle Ophthalmic Solution (Placebo Comparator): Placebo Ophthalmic Solution
  Interventions: Drug: Placebo Ophthalmic Solution

INTERVENTIONS:
Drug: 1% Tavilermide Ophthalmic Solution — 1% Tavilermide BID Dosing
  Arms: Tavilermide Ophthalmic Solution
Drug: Placebo Ophthalmic Solution — Vehicle Ophthalmic Solution
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Tavilermide Ophthalmic Solution compared with Placebo Ophthalmic Solution in treating the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

Be at least 18 years of age Provided written informed consent Have a reported history of dry eye Have a history of use or desire to use eye drops for dry eye

Exclusion Criteria:

Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation (e.g. follicular conjunctivitis) at Visit 1, or have been diagnosed with ocular rosacea, or any viral or bacterial disease of the cornea or conjunctiva, within the last 12 months Have any planned ocular and/or lid surgeries over the study period Have corrected visual acuity greater than or equal to +0.7 as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in both eyes at Visit 1 Have an uncontrolled systemic disease Be a woman who is pregnant, nursing or planning a pregnancy Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; IUD; or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use adequate birth control as defined above for the remainder of the study Have a known allergy and/or sensitivity to the test article or its components Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 45 days of Visit 1 Be unable or unwilling to follow instructions, including participation in all study assessments and visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2015-12; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Corneal Fluorescein Staining | Day 57
Ocular Discomfort | Day 57

SECONDARY OUTCOMES:
Corneal Fluorescein Staining | Day 15
Ocular Surface Disease Index | Day 57
Ocular Dryness | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Garth Cumberlidge, PhD, Study Director — Mimetogen Pharmaceuticals USA, Inc.
Locations (2):
- United States (2):
  - MIM-727 Investigational Site, Louisville, Kentucky
  - MIM-727 Investigational Site, Nashville, Tennessee